CLINICAL TRIAL: NCT00086034
Title: Phase II Trial of Motexafin Gadolinium (MGd) in Patients With Relapsed or Refractory Indolent Non-Hodgkin's Lymphoma
Brief Title: Study of Motexafin Gadolinium for the Treatment of Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-0221
Record Dates: First submitted 2004-06-21; First posted 2004-06-23 (Estimated); Last update posted 2007-05-15 (Estimated); Status verified 2007-05

CONDITIONS: Lymphoma; Non-Hodgkin's Lymphoma
Keywords: Lymphoma; Non-Hodgkin's Lymphoma; Indolent lymphoma; Relapsed lymphoma; Refractory lymphoma; Motexafin gadolinium
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin | interventions — motexafin gadolinium

INTERVENTIONS:
Drug: Motexafin gadolinium

SUMMARY:
The primary purpose of this study is to find out if motexafin gadolinium may be an effective treatment for patients with non-Hodgkin's lymphoma (NHL). Secondly, the safety and side effects of motexafin gadolinium will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Refractory or relapsed indolent NHL. Eligible WHO histologies include follicular NHL (Grades 1, 2, and 3); marginal zone nodal; marginal zone splenic; and mucosa-associated lymphoid tissue (MALT) types
* Failed ≥ 1 previous regimens, one of which must have contained rituximab as either a single agent or in combination with chemotherapy
* ECOG performance status score either 0 or 1
* Willing and able to provide written informed consent

Exclusion Criteria:

Laboratory values of:

* Platelet count < 50,000/µL
* AST or ALT > 2 x the upper limit of normal (ULN)
* Total bilirubin > 2 x ULN
* Creatinine > 2.0 mg/dL

and

* Greater than three prior regimens (where a regimen is defined as a treatment for NHL given after disease progression)
* Uncontrolled hypertension
* Known history of porphyria, G6PD deficiency, HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35

PRIMARY OUTCOMES:
Clinical response rate

SECONDARY OUTCOMES:
Progression-free survival
Duration of clinical response
Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Brad Kahl, MD, Principal Investigator — University of Wisconsin, Madison
Locations (7):
- United States (7):
  - San Diego, California
  - Stanford, California
  - Miami, Florida
  - Chicago, Illinois
  - Baltimore, Maryland
  - Rochester, Minnesota
  - Madison, Wisconsin